CLINICAL TRIAL: NCT03257007
Title: Mindfulness to Enhance Quality of Life and Support Advance Care Planning (MEANING): A Randomized Controlled Pilot Trial for Adults With Metastatic Cancer and Their Family Caregivers
Brief Title: Mindfulness to Enhance Quality of Life and Support Advance Care Planning
Acronym: MEANING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Shelley Johns, Assistant Professor of Medicine, Research Scientist, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1702223546
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Mindfulness; Meditation; Metastatic Cancer; Quality of Life; Advance Care Planning; Palliative Care; Family Caregiver; Supportive Care
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Participants will be assigned in equal numbers using block randomization to the mindfulness intervention or usual care. The course curriculum for the mindfulness intervention is modeled on the Mindfulness-Based Stress Reduction program which involves intensive experiential training of participants in secular mindfulness meditation practices (i.e., body scan, sitting meditation, gentle hatha yoga with chair adaptations, compassion meditation), with an emphasis on embodying interpersonal mindfulness in dialogue.
Masking Description: Participants are blind to study hypotheses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants assigned to Usual Care will continue to receive standard care from their oncology team, including access to supportive care from oncology social workers. At the end of the study, usual care dyads will receive a packet of informational materials on mindfulness meditation, receive a CD with 5 mindfulness meditation practices, and meet with the study interventionist for guidance on how to use the materials and mindfulness recordings to their advantage in coping with cancer-related challenges.
- Mindfulness (Active Comparator): The Mindfulness intervention will consist of six 2-hour sessions that will include guided mindfulness practices, didactics, and group discussion. The course curriculum is modeled on the Mindfulness-Based Stress Reduction program which involves intensive experiential training of participants in secular mindfulness meditation practices (i.e., body scan, sitting meditation, gentle hatha yoga with chair adaptations, compassion meditation), with an emphasis on embodying interpersonal mindfulness in dialogue.
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — The Mindfulness intervention sessions are designed to cultivate present-moment awareness in everyday life to facilitate adaptive and non-reactive relating to thoughts, feelings, and bodily sensations. Participants will be provided with 10-20 minute audio recordings of each of 5 mindfulness practices covered in class, recorded in the facilitator's voice. Participants will be encouraged to practice mindfulness at home 10-20 minutes per day, 6 days per week. Participants will be provided with weekly diaries on which to record type and amount of home practice of mindfulness skills.
  Arms: Mindfulness

SUMMARY:
The MEANING trial is a randomized controlled mixed methods pilot designed to compare a novel mindfulness meditation-based intervention (MEANING) to usual care for adults with advanced-stage solid malignancies and their family caregivers.

DETAILED DESCRIPTION:
Mindfulness meditation practices have reduced emotional distress, avoidant coping, and improved spiritual well-being in adult cancer patients. These beneficial effects may occur through present-moment acceptance of unpleasant thoughts, feelings, and circumstances and adaptive coping through self-awareness, self-regulation, and self-transcendence. Most mindfulness trials in cancer have focused on early-stage survivors; however, preliminary evidence suggests that mindfulness may help reduce distress in patients with advanced cancer and their family caregivers (FCGs).

Sixty patients with an advanced-stage solid malignancy and their FCGs (60 dyads) will be randomized in equal numbers to receive either the 6-week mindfulness intervention or usual care. Both groups will receive standard cancer care throughout the study period. Dyads randomized to the mindfulness arm will learn mindfulness meditation practices (e.g., body scan, sitting meditation) and mindful communication practices to enhance quality of life, support advance care planning engagement, and improve a variety of secondary outcomes.

The study will use a mixed methods 2-arm randomized design to examine the effects of the mindfulness intervention compared to usual care and seek to explain trial results using insights gleaned from post-intervention qualitative interviews.

ELIGIBILITY:
Inclusion Criteria-Patients

* Patient is at least 18 years of age.
* Patient is at least 3 weeks post-diagnosis of an incurable (locally advanced or metastatic) solid malignancy.
* Patient's attending medical oncologist would not be surprised if the patient died in the next 12 months.
* Patient has not completed a POST form.
* Patient scores ≥ 7 on the Mini-Mental Adjustment to Cancer cognitive avoidance subscale.
* Patient is willing and able to consent and travel to the class location for 6 weekly 2-hour sessions.
* Patient has a family member or close friend eligible and interested in participating in the study.
* Patient has adequate English fluency for completion of data collection

Inclusion Criteria-Family Care Givers (FCG)

* FCG is at least 18 years of age.
* FCG has been invited to participate in the trial with a patient who meets eligibility criteria above.
* FCG is willing and able to consent and travel to the class location for 6 weekly 2-hour sessions.
* FCG has adequate English fluency for completion of data collection

Exclusion Criteria-Patients

* Patient reports a score of > 2 on the Activities and Function item from the Patient Generated Subjective Global Assessment91 (PG-SGA; the patient-reported version of the Eastern Cooperative Oncology Group score).
* Patient makes 3 or more errors on a validated 6-item cognitive screener or exhibits significant psychiatric or cognitive impairment (e.g., dementia/delirium, retardation, active psychosis) that in the judgment of the investigators would preclude providing informed consent and study participation.
* Currently receiving hospice care (patients who enroll in hospice during the trial will have the option of continuing trial participation).

Exclusion Criteria-FCGs

• FCG exhibits significant psychiatric or cognitive impairment (e.g., dementia/delirium, retardation, active psychosis) that in the judgment of the investigators would preclude providing informed consent and study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in quality of life (QoL) for Patients | Baseline, 6 weeks, and 10 weeks
  QoL for patients will be assessed with the McGill Quality of Life Inventory.
Change from baseline in quality of life (QoL) for Family Caregivers | Baseline, 6 weeks, and 10 weeks
  QoL for family caregivers will be assessed with the Caregiver Quality of Life - Cancer scale (CQoLC).

SECONDARY OUTCOMES:
Change from baseline in advance care planning (ACP) stage of change | Baseline, 6 weeks, and 10 weeks
  ACP stage of change will be assessed by a measure modified from Fried et. al assessing stage of change for 3 advance care planning behaviors (completing a living will, medical power of attorney form, or POLST form; patient only measure).
Change from baseline in advance care planning (ACP) engagement | Baseline, 6 weeks, and 10 weeks
  ACP engagement (self-efficacy, readiness) will be measured using 2 subscales of the Advance Care Planning Engagement Survey (patient only measure).
Change from baseline in caregiver burden | Baseline, 6 weeks, and 10 weeks
  Caregiver burden will be measured using the Zarit Burden Interview (family caregiver measure only)
Change from baseline in avoidant coping | Baseline, 6 weeks, and 10 weeks
  Avoidant coping will be assessed using the Mini-MAC Cognitive Avoidance subscale
Change from baseline in avoidant coping | Baseline, 6 weeks, and 10 weeks
  Avoidant coping will be assessed using the Brief COPE Self-Distraction, Denial, and Behavioral Disengagement subscales
Change from baseline in depressive symptoms | Baseline, 6 weeks, and 10 weeks
  Depressive symptoms will be assessed using the PHQ-8
Change from baseline in anxiety | Baseline, 6 weeks, and 10 weeks
  Anxiety will be assessed using the GAD-7
Change from baseline in spiritual well-being | Baseline, 6 weeks, and 10 weeks
  Spiritual well-being will be measured using the FACIT-SP.
Change from baseline in sleep disturbance | Baseline, 6 weeks, and 10 weeks
  Sleep disturbance will be assessed using the PROMIS Sleep Disturbance.
Change from baseline in family communication | Baseline, 6 weeks, and 10 weeks
  Family communication will be assessed using the Social Constraint Scale
Change from baseline in interpersonal closeness | Baseline, 6 weeks, and 10 weeks
  Interpersonal closeness will be assessed using the Perceived Interpersonal Closeness Scale.
Change from baseline in acceptance of illness | Baseline, 6 weeks, and 10 weeks
  Acceptance of illness will be assessed using the PEACE Scale.
Change from baseline in mindfulness | Baseline, 6 weeks, and 10 weeks
  Mindfulness will be assessed using the FFMQ-SF Non-reactivity to Internal Experience and Acting with Awareness subscales.
Distress Thermometer | Baseline, 6 weeks, and 10 weeks
  Distress will be assessed using the Distress Thermometer.
Intervention satisfaction and helpfulness | 6 weeks
  Satisfaction and helpfulness with the Mindfulness intervention will be assessed using single-item investigator-created 7- and 10-point Likert scales, respectively (Mindfulness group only).

CONTACTS AND LOCATIONS:
Overall Officials: Shelley A Johns, PsyD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mosher CE, Beck-Coon KA, Wu W, Lewson AB, Stutz PV, Brown LF, Tang Q, Helft PR, Levoy K, Hickman SE, Johns SA. Mindfulness to enhance quality of life and support advance care planning: a pilot randomized controlled trial for adults with advanced cancer and their family caregivers. BMC Palliat Care. 2024 Sep 28;23(1):232. doi: 10.1186/s12904-024-01564-7. PMID 39342143

DOCUMENTS (1):
  • Informed Consent Form (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT03257007/ICF_000.pdf